CLINICAL TRIAL: NCT03891771
Title: Seniors Guardian: A Non-intrusive Monitoring Platform for Activities of Daily Living Amongst the Elderly
Brief Title: Seniors Guardian: A Monitoring Platform for the Elderly
Acronym: SEMONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Servicio de Vivienda y Urbanismo, Chile (Unknown); Ilustre Municipalidad de San Antonio, Chile (Unknown); Corporación Municipal de Valparaíso, Chile (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CEC181-18
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Quality of Life
Keywords: Elderly; Activities of daily living; Telemonitoring

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients allocated to usual care will receive standard follow-up procedures at their primary care facility.
- Telemonitoring sensors (Experimental): Patients allocated to this arm will receive a complex sensor platform aimed at detecting falls at home, nocturia and several environmental variables, including carbon monoxide concentrations, humidity and temperature. The system also includes a panic button that can be used to request assistance in emergencies.
  Interventions: Device: Telemonitoring sensors

INTERVENTIONS:
Device: Telemonitoring sensors — This complex platform entails several sensors aimed at detecting falls, nocturia and environmental variables in the participant's home. Sensors are non-intrusive and its only wearable component is the panic button which must be carried by the participant.
  Arms: Telemonitoring sensors

SUMMARY:
This pilot study evaluates whether a telemonitoring platform of activities of daily living amongst the elderly can improve their quality of life. Participants will be randomised to two different follow-up strategies, one comprising a monitoring platform and the other standard visits at a healthcare facility. Quality of life will be assessed using standardised questionnaires.

DETAILED DESCRIPTION:
Elderly participants at perceived socioeconomic risk will be randomised in a 1:1 ratio to receive either a telemonitoring platform in their houses or standard health care. The platform will include sensors able to detect falls, nocturia (which have been previously validated) and sensors for environmental variables including humidity, carbon monoxide levels and temperature. In addition, a wearable panic button will be provided for participants allocated to the sensor platform which will allow them to obtain help in case of an emergency. The sensor platform will be connected to emergency services and healthcare providers,and they should receive and react to any anomaly detected in their readings.

Participants will be followed up for 10 months. Quality of life questionnaires, including the World Health Organisation's WHOQOL-BREF and the EQ-5D for health-related quality of life, will be used to address potential intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Elderly participant (>65 years of age) perceived to be at socioeconomic risk
* Resident in the city of Valparaiso or San Antonio
* Lives alone
* Obtained a housing subsidy from the Servicio de Vivienda y Urbanismo (Housing and Urbanism Services)

Exclusion Criteria:

* Dementia
* Substance or alcohol abuse
* Inability to answer quality of life questionnaires due to medical or psychiatric morbidity
* Terminal illness (life expectancy under 6 months)
* Ownership of pets within the residence (ie. dogs, cats).
* Refusal to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Overall Quality of Life score as measured by the World Health Organisation Quality of Life Questionnaire (WHOQOL-BREF) | 1 month after randomisation
  This scale is designed to assess the overall quality of life of the respondent using 5-point Likert scales. Higher scores mean a better quality of life. WHOQOL-BREF is divided in 4 domains, including physical health, psychological, social relationships and environment. The mean score for each domain is used to calculate the domain score. Scores can then be added together to obtain an overall score. Therefore, scores in the WHOQOL-BREF questionnaire range from 4 to 20 points.
Overall Quality of Life score as measured by the World Health Organisation Quality of Life Questionnaire (WHOQOL-BREF) | 5 months after randomisation
  This scale is designed to assess the overall quality of life of the respondent using 5-point Likert scales. Higher scores mean a better quality of life. WHOQOL-BREF is divided in 4 domains, including physical health, psychological, social relationships and environment. The mean score for each domain is used to calculate the domain score. Scores can then be added together to obtain an overall score. Therefore, scores in the WHOQOL-BREF questionnaire range from 4 to 20 points.
Overall Quality of Life score as measured by the World Health Organisation Quality of Life Questionnaire (WHOQOL-BREF) | 10 months after randomisation
  This scale is designed to assess the overall quality of life of the respondent using 5-point Likert scales. Higher scores mean a better quality of life. WHOQOL-BREF is divided in 4 domains, including physical health, psychological, social relationships and environment. The mean score for each domain is used to calculate the domain score. Scores can then be added together to obtain an overall score. Therefore, scores in the WHOQOL-BREF questionnaire range from 4 to 20 points.
Health-Related Quality of Life score using the EuroQOL-5D (EQ-5D) Questionnaire | 1 month after randomisation
  EuroQol-5D (EQ-5D) is a standardised questionnaire that allows to quantify health-related quality of life. It is divided in two sections, a descriptive section and a visual analogue scale (VAS) at the end of the questionnaire. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-VAS records the patient's self-rated health on a vertical visual analogue scale. Results are presented as a descriptive profile or as an index value calculated from the descriptive component which is country-specific. Visual analog values can range from 0 to 100, with higher values indicating an overall better health-related quality of life.
Health-Related Quality of Life score using the EuroQOL-5D (EQ-5D) Questionnaire | 5 months after randomisation
  EuroQol-5D (EQ-5D) is a standardised questionnaire that allows to quantify health-related quality of life. It is divided in two sections, a descriptive section and a visual analogue scale (VAS) at the end of the questionnaire. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-VAS records the patient's self-rated health on a vertical visual analogue scale. Results are presented as a descriptive profile or as an index value calculated from the descriptive component which is country-specific. Visual analog values can range from 0 to 100, with higher values indicating an overall better health-related quality of life.
Health-Related Quality of Life score using the EuroQOL-5D (EQ-5D) Questionnaire | 10 months after randomisation
  EuroQol-5D (EQ-5D) is a standardised questionnaire that allows to quantify health-related quality of life. It is divided in two sections, a descriptive section and a visual analogue scale (VAS) at the end of the questionnaire. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-VAS records the patient's self-rated health on a vertical visual analogue scale. Results are presented as a descriptive profile or as an index value calculated from the descriptive component which is country-specific. Visual analog values can range from 0 to 100, with higher values indicating an overall better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Taramasco, Ph.D., Study Chair — Universidad de Valparaiso; Felipe T Martinez, M.D., M.Sc, Principal Investigator — Universidad Andres Bello
Locations (4):
- Chile (4):
  - Centro de Salud Familiar 30 de Marzo, San Antonio
  - Centro de Salud Familiar Barrancas, San Antonio
  - Centro de Salud Familiar Nestor Fernandez, San Antonio
  - Centro de Salud Familiar San Antonio, San Antonio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson BE, Barry PP, Renick N, Bergen MR, Stratos GA. Physician confidence and interest in learning more about common geriatric topics: a needs assessment. J Am Geriatr Soc. 2001 Jul;49(7):963-7. doi: 10.1046/j.1532-5415.2001.49188.x. PMID 11527489
- [Background] Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P; CONSORT Group. Methods and processes of the CONSORT Group: example of an extension for trials assessing nonpharmacologic treatments. Ann Intern Med. 2008 Feb 19;148(4):W60-6. doi: 10.7326/0003-4819-148-4-200802190-00008-w1. PMID 18283201
- [Background] Stoddart A, Hanley J, Wild S, Pagliari C, Paterson M, Lewis S, Sheikh A, Krishan A, Padfield P, McKinstry B. Telemonitoring-based service redesign for the management of uncontrolled hypertension (HITS): cost and cost-effectiveness analysis of a randomised controlled trial. BMJ Open. 2013 May 28;3(5):e002681. doi: 10.1136/bmjopen-2013-002681. PMID 23793650
- [Background] Lewis KE, Annandale JA, Warm DL, Hurlin C, Lewis MJ, Lewis L. Home telemonitoring and quality of life in stable, optimised chronic obstructive pulmonary disease. J Telemed Telecare. 2010;16(5):253-9. doi: 10.1258/jtt.2009.090907. Epub 2010 May 18. PMID 20483881
- See also: Home telemonitoring or structured telephone support programmes after recent discharge in patients with heart failure : systematic review and economic evaluation Scientific summary — https://www.ncbi.nlm.nih.gov/books/NBK260871/
- See also: Espinoza I, Osorio P, Torrejón MJ, Lucas-Carrasco R, Bunout D. Validación del cuestionario de calidad de vida (WHOQOL-BREF) en adultos mayores chilenos. Rev Med Chile [Internet]. 2011;579-86 — http://www.scielo.cl/pdf/rmc/v139n5/art03.pdf